CLINICAL TRIAL: NCT07202650
Title: EFFECT OF GUIDED IMAGERY ON PREMENSIVE SYNDROME IN UNIVERSITY STUDENTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KA24/415
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Guided Imagery
Keywords: Premenstrual syndrome, guided imagery, quality of life
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): At baseline, students in both the intervention and control groups will complete the Introductory Characteristics Data Collection Form, the Premenstrual Syndrome Scale, and the WHO Quality of Life Scale. Students in the intervention group with high PMS scores will be instructed to practice guided imagery for 15 minutes daily during two consecutive menstrual cycles-specifically, during the seven days prior to menstruation when symptoms begin and the first four days of menstruation. The control group will receive no intervention.
  Throughout the study, intervention group participants will complete the Menstrual Cycle Follow-up Form and the Guided Imagery Follow-up Form, while control group participants will complete only the Menstrual Cycle Follow-up Form. After two cycles, both groups will again complete the Premenstrual Syndrome Scale and the WHO Quality of Life Scale.
  Interventions: Behavioral: guided imagery
- control group (No Intervention): At baseline, students in both the intervention and control groups will complete the Introductory Characteristics Data Collection Form, the Premenstrual Syndrome Scale, and the WHO Quality of Life Scale. No intervention will be applied to the control group; however, they will be asked to complete the Menstrual Cycle Follow-up Form throughout the study. After two menstrual cycles, both groups will again complete the Premenstrual Syndrome Scale and the WHO Quality of Life Scale.

INTERVENTIONS:
Behavioral: guided imagery — Guided imagery is a form of mind-body communication, defined as a flow of thoughts involving what we smell, taste, see, hear, and touch, or as the way the mind encodes, stores, and retrieves information. Guided imagery is based on the understanding that the mind and body are interconnected and that the mind can influence bodily functions. Stress and anxiety directly affect the brain and the immune system.
  Arms: intervention group

SUMMARY:
Premenstrual Syndrome (PMS) is typically defined as a condition characterized by physical, behavioral, and emotional symptoms that typically appear at the end of the luteal phase of the menstrual cycle, occur 7-10 days before menstruation, and disappear at the onset of menstruation or shortly thereafter.

The symptoms of PMS include irritability, a feeling of losing control, anxiety, depression, insomnia, hypersomnia, decreased concentration, and unexplained crying. Symptoms of PMS include irritability, a sense of losing control, anxiety, depression, insomnia, hypersomnia, decreased concentration, unexplained crying, fatigue, weakness, increased appetite, edema, weight gain, dizziness, headaches, joint pain, muscle pain, mastalgia, breast tenderness, aggressiveness, decreased or increased sexual activity, and avoidance of social interactions. Studies have also shown that premenstrual symptoms in young women negatively affect their self-confidence, social relationships, quality of life, and academic performance. For this reason, PMS treatment is important. PMS treatment focuses on alleviating physical and psychiatric symptoms. In PMS treatment, various dietary supplements and complementary-alternative methods can be utilized.

Alternative and complementary therapies such as reflexology, pilates, acupressure, music, exercise, and guided imagery have shown promising results in reducing premenstrual symptoms. PMS treatment can be approached from multiple angles. It is important to address the underlying causes of PMS and to consider the individual's overall well-being.It is known that mind-body-based approaches in complementary and alternative medicine have a healing effect on individuals from a psychological perspective. Guided imagery is a form of mind-body communication and is defined as a stream of thoughts or the way in which our minds encode, store, and express information based on what we smell, taste, see, hear, and touch. Guided imagery is based on the understanding that the body and mind are interconnected and that the mind can influence the body. Guided imagery has been found to be effective in various situations, such as reducing stress, improving mood, strengthening the immune system, reducing fatigue, improving sleep quality, and minimizing nausea and vomiting. There are very few studies in the literature on the use of guided imagery to reduce symptoms in university students during the premenstrual period. The aim of this study is to investigate the effect of guided imagery on premenstrual syndrome in university students.

DETAILED DESCRIPTION:
Premenstrual Syndrome (PMS) is defined as a condition characterized by physical, behavioral and emotional symptoms that typically occur at the end of the luteal phase of a woman's menstrual cycle and occur 7- 10 days before menstruation, disappear at the onset of menstruation or shortly after (Chumpalova et al.Premenstrual Syndrome (PMS) is defined as a condition characterized by physical, behavioral and emotional symptoms that typically occur at the end of the luteal phase of a woman's menstrual cycle and occur 7- 10 days before menstruation, disappear at the onset of menstruation or shortly after (Chumpalova et al., 2007).When diagnosing PMS, a symptom diary should be kept by a woman for at least 2 menstrual cycles. The entries in the diary should describe the symptoms that occur during the luteal phase, which ends with the onset of menstruation, and the subsequent symptom-free week until ovulation.he entries in the diary should describe the symptoms that occur during the luteal phase, which ends with the onset of menstruation, and the entries in the diary should describe the symptoms that occur during the luteal phase, which ends with the onset of menstruation, and the subsequent symptom-free week until ovulation. Underlying physical or psychological disorders that may cause symptom exacerbation should be ruled out (Gnanasambanthan and Datta, 2022). According to The American College of Obstetricians and Gynecologists (ACOG), according to the American Society of Obstetrics and Gynecology, a woman's symptoms can be diagnosed with PMS; for at least three menstrual cycles in a row, it should be within five days before menstruation, end within four days after menstruation begins, and prevent some normal activities (ACOG, 2023).or at least three menstrual cycles in a row, it should be within five days before menstruation, end within four days after menstruation begins, and prevent some normal activities (ACOG, 2023). According to the Association of Women's Health, Obstetric and Neonatal Nurses (AWHONN), factors such as medical, psychological, sociocultural and lifestyle should be taken into account when evaluating PMS (AWHONN, 2003). Symptoms of PMS include irritability, feeling of losing control, anxiety, depression, insomnia, hypersomnia, Dec Novation of concentration, crying for no reason, weakness, fatigue, increased appetite, edema, weight gain, dizziness, headache, joint pain, muscle pain, mastalgia, fullness of breasts, tendency to fight, decrease or increase in sexual activity, avoidance of social relationships, such as more than 200 different psychological, physical and behavioral symptoms (Silva et al.Symptoms of PMS include irritability, feeling of losing control, anxiety, depression, insomnia, hypersomnia, Dec Novation of concentration, crying for no reason, weakness, fatigue, increased appetite, edema, weight gain, dizziness, headache, joint pain, muscle pain, mastalgia, fullness of breasts, tendency to fight, decrease or increase in sexual activity, avoidance of social relationships, such as more than 200 different psychological, physical and behavioral symptoms (Silva et al.,2006).

Up to 90% of women of childbearing age report that they perceive one or more symptoms in the days before menstruation; these symptoms can change their behavior and well-being and therefore affect their family, social and business environment (Campagne et al.p to 90% of women of childbearing age report that they perceive one or more symptoms in the days before menstruation; these symptoms can change their behavior and well-being and therefore affect their family, social and business environment (Campagne et al.,2007; Freeman, 2003). Although the etiology of PMS is not known for sure, it is believed that endocrine factors such as carbohydrate intolerance, fluid retention, progesterone deficiency, estrogen deficiency or excess, endogenous endorphins deficiency, renangiotensin and aldosterone imbalance, adrenal gland hyperactivity, central catecholamine imbalance, thyroid dysfunction, hyperprolactinemia, hypoglycemia, as well as psychological factors such as genetic factors and stress are effective in its development ( According to Amjadian et al.Although the etiology of PMS is not known for sure, it is believed that endocrine factors such as carbohydrate intolerance, fluid retention, progesterone deficiency, estrogen deficiency or excess, endogenous endorphins deficiency, renangiotensin and aldosterone imbalance, adrenal gland hyperactivity, central catecholamine imbalance, thyroid dysfunction, hyperprolactinemia, hypoglycemia, as well as psychological factors such as genetic factors and stress are effective in its development ( According to Amjadian et al.,2022).

Traditionally considered a concern among women of childbearing age, PMS is rapidly becoming a common mental illness, significantly impairing many women's ability to function on a daily basis (Erbil et al.,2023)raditionally considered a concern among women of childbearing age, PMS is rapidly becoming a common mental illness, significantly impairing maditionally considered a among women of childbearing age, PMS is rapidly becoming a common mental illness, significantly impairing many women's ability to function on a daily basis (Erbil et al.,2023). Meanwhile, in the context of the COVID-19 pandemic, there has been an increase in the incidence of some symptoms in PMS( Aolymat et al., 2022). A review of gynecological disease burden data in China highlights PMS as one of the top three gynecological diseases affecting women aged 15 to 49 (Ji et al., 20016). Due to the variety of PMS symptoms, it is quite difficult to determine and evaluate the true prevalence of PMS (Topatan and Kahraman, 2020).ue to the variety of PMS symptoms, it is quite difficult to determine and evaluate the true prevalence of PMS (Topatan and Kahraman, 2020). StDue to the variety of PMS symptoms, it is quite difficult to determine and evaluate the true prevalence of PMS (Topatan and Kahraman, 2020). Studies conducted around the world report that the prevalence of PMS varies between 7.1% and 99.5% ( Eshetu et al., 2022; Yi et al.,2023; Yang et al.,2024).It is observed that the frequency of PMS varies between 36.3-91.8% in studies involving university students in our country (Bakır and Beji, 2021; Karaküçük et Dec.,2022; Afacan and Kabakci,2023) Studies have shown that women use both pharmacological and non-pharmacological strategies to manage physical and psychological symptoms during the premenstrual period (Sehati-Shafaie et al.facan and Kabakci,2023) Studies have shown that women use both pharmacological and non-pharmacological strategies to manage physical and psychological symptoms during the premenstrual period (Sehati-Shafaie et al.,2018; Jebakani,2019). StAfacan and Kabakci,2023) Studies have shown that women use both pharmacological and non-pharmacological strategies to manage physical and psychological symptoms during the premenstrual period (Sehati-Shafaie et al.,2018; Jebakani,2019). Studies have also shown that young women with premenstrual symptoms have a negative impact on their self-confidence, social relationships, quality of life and academic achievement of students (Farrokh-Eslamlou et al., 2015; Behboudi-Gandevani et al., 2017; Nakame et al., 2019, Nyirenda et al.,2023;Esan et al., 2024). Therefore, PMS treatment is gaining importanceakame et al., 2019, Nyirenda et al.,2023;Esan et al., 2024). Therefore, PMS treatment is gaining importance. PMS treatment focuses on relieving physical and psychiatric symptoms. Various food suppleakame et al., 2019, Nyirenda et al.,2023;Esan et al., 2024). Therefore, PMS treatment is gaining importance. PMS treatment focuses on relieving physical and psychiatric symptoms. Various food supplements and complementary-alternatiNakame et al., 2019, Nyirenda et al.,2023;Esan et al., 2024). Therefore, PMS treatment is gaining importance. PMS treatment focuses on relieving physical and psychiatric symptoms. Various food supplements and complementary-alternative methods can be used in the treatment of PMS (Hofmeister and Bodden, 2016). Internative and complementary therapies such as reflexology, pilates, acupressure, music, exercise and directed imagery have shown promising results in reducing premenstrual symptoms (Groer and Ohnesorge, 1993; Bazarganipour et al.,2017; According to Askari et al.,2018).It is known that mind-body based approaches in complementary and alternative medicine applications have a healing effect on individuals from a psychological point of view (Bulduklu, 2015).ccording to Askari et al.,2018).It is known that mind-body based approaches in complementary and alternative medicine applications have a healing effect on individuals from a psychological point of view (Bulduklu, 2015). The most commonly used technique in mind-body based applications is "relaxation" and thccording to Askari et al.,2018).It is known that mind-body based approaches in complementary and alternative medicine applications have a healing effect on individuals from a psychological point of view (Bulduklu, 2015). The most commonly used technique in mind-body based applications is "relaxation" and the main purpose of this relaxation technique is to neutralize stress-related physical changes, for example November muscle density, high blood pressure and hormone changes, while calming the mind (Coats and Feldman, 2011). Directed imagery; It is a way of mind-body communication and is basically defined as a flow of thoughts or the way our mind encodes, stores and reveals information that we smell, taste, see, hear and touch.t is a way of mind-body communication and is basically defined as a flow of thoughts or the way our mind encodes, stores and reveals information that we smell, taste, see, hear and touch. Directed imagery is based on the understanding that the body and the mind are connected and that the mind can influence the body. Stress and anxiety directly affect the brain and the immune system (Roffe et al., 2005).

It can be practiced either through an instructor actively guiding the person or by listening to an audio or video recording prepared by an instructor and played back to the person. The person can practice self-directed imagery without the need for an outsidet can be practiced either through an instructor actively guiding the person or by listening to an audio or video recording prepared by an instructor and played back to the person. The person can practice self-directed imagery without the need for an outside instructor. A person can create his own scenario. The method can be applied in groups, as well as it is possible to make one-on-one application. Directed imagery has been found effective in various situations such as reducing stress, improving mood, strengthening the immune system, reducing fatigue, improving sleep quality, minimizing nausea and vomiting (Trakhtenberg, 2008; Yoo et al.Directed imagery has been found effective Directed imagery has been found effective in various situations such as reducing stress, improving mood, strengthening the immIn a study conducted by Patel (2017) among university students, when the effectiveness of directed imagery technique in alleviating premenstrual syndrome was evaluated, it was found that directed imagery reduces premenstrual symptoms (Patel, 2017).n a study conducted by Patel (2017) among university students, when the effectiveness of directed imagery technique in alleviating premenstrual syndrome was evaluated, it was found that directed imagery reduces premenstrual symptoms (Patel, 2017). In a study conducted by Heydarpur and Dehghan (2019), it was found that premenstrual syndrome was alleviated in university students by comparing the effectiveness of hypnotherapy and virtual reality technology relaxation in alleviating the symptoms of premenstrual syndrome (Heydarpur and Dehghan, 2019). In the literature, studies in which directed imagery was performed to reduce symptoms during the premenstrual period in university students are quite limited.

The Hypothesis of the StudyIn the literature, studies in which directed imagery was performed to reduce symptoms during the premenstrual period in university students are quite limited.

ELIGIBILITY:
Inclusion Criteria:

* Regular menstrual cycles (21-35 days over the last three cycles)

Age 18 years or older

No medical treatment for PMS

Ability to communicate effectively in Turkish

No psychiatric diagnosis or gynecological disorder (e.g., abnormal uterine bleeding, myoma, ovarian cysts)

A score >89 on the Premenstrual Syndrome Scale (PMSS)

No prior participation in guided imagery training

Exclusion Criteria:

* Failure to perform guided imagery at the correct time or in the prescribed manner

Irregular menstruation during the last three months

Use of contraceptives

Use of analgesics during menstruation while participating in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women participants
Enrollment: 48 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
premenstrual syndrome | two months
  The Premenstrual Syndrome Scale, developed by Gençdoğan (2006), is a five-point Likert-type instrument consisting of 44 items designed to assess the severity of premenstrual symptoms, based on DSM-III and DSM-IV-R criteria. In scoring, responses are rated as follows: "None" = 1 point, "Very little" = 2 points, "Sometimes" = 3 points, "Often" = 4 points, and "Always" = 5 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Başkent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No